CLINICAL TRIAL: NCT06377709
Title: A Mixed-methods Acceptability Study of ProACTive, an Early Acceptance and Commitment Therapy Intervention to Help Burns Patients Adjust to Changes to Appearance
Brief Title: A Mixed-methods Acceptability Study of ProACTive to Help Burns Patients Adjust to Changes to Appearance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 24CP001
Record Dates: First submitted 2024-04-17; First posted 2024-04-22 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Burn Injuries; Burns; Emotional Distress; Adjustment
MeSH Terms: conditions — Burns | interventions — Coping Skills

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ProACTive intervention (Experimental): ProACTive intervention. Participants will choose how many, and which, modules to complete.
  Interventions: Other: ProACTive

INTERVENTIONS:
Other: ProACTive — ProACTive intervention, a talking therapy utilising acceptance and commitment therapy (ACT) techniques.

SUMMARY:
This mixed-methods acceptability study aims to investigate whether an early acceptance and commitment therapy (ACT) based intervention called ProACTive, aimed at supporting burns patients' adjustment to a changed appearance and preventing distress, is acceptable. This will be measured by descriptive data, questionnaire data and semi-structured interviews.

Preliminary data on the potential clinical effectiveness of the intervention will also be gathered. This will be measured by scores on standardised questionnaires.

DETAILED DESCRIPTION:
Evidence suggests that appearance concerns after burn injuries start early. Appearance concerns can be chronic, create psychological distress and impact quality of life. No early psychological interventions for appearance concerns after burn injuries currently exist.

ProACTive, a novel psychological intervention (talking therapy), utilising acceptance and commitment therapy (ACT) techniques with an additional focus on developing self-compassion and social skills training, was developed. It aims to help burns patients adjust to changes to appearance and prevent distress. It involves up to five 30-minute modules and patients can select how many, and which, modules to complete. It is delivered by a psychological professional working in burns services.

The primary aim of this study is to explore whether the ProACTive intervention is acceptable to burns patients. A secondary objective is to gather preliminary data on the potential clinical effectiveness of the ProACTive intervention.

A mixed-methods single-arm acceptability study will be conducted.

ProACTive will be offered to burns patients (aged 18 years or over) meeting inclusion criteria and admitted to the burns service at Nottingham University Hospitals NHS Trust.

Fifteen participants will be recruited to complete the intervention.

The primary objective of exploring the acceptability of the ProACTive intervention will be measured by:

* Intervention update rate (percentage of those invited to participate in the study)
* Descriptive data about reasons for not taking up the intervention (if patients consent to participating in the study in this way)
* Patient feedback gathered through a semi-structured exit interview as soon as possible after the intervention ends (within two weeks)
* Patient feedback gathered using a standardised self-report questionnaire to record helpful and hindering aspects of the intervention will be completed after every session completed.
* Descriptive data about how many, and which of, the sessions patients choose to complete and the spacing of sessions completed
* The number of sessions completed during hospital admission and after hospital discharge, and whether these were completed face to face or virtually
* Descriptive data about participants' preferences for receiving the post-session resources in paper or electronic format
* The number of times participants viewed the post-session online videos containing audio-exercises
* Descriptive data about reason for ending the intervention before all sessions have been completed

Template analysis (King, 2012), a form of thematic analysis (Braun & Clarke, 2006), will be used to analyse patterns of meaning, or themes, within the transcripts of the interviews. The Theoretical Framework of Acceptability (TFA; Sekhon et al., 2017) will also be used to develop the interview schedule and the initial coding template.

The secondary objective to gather preliminary data on the potential clinical effectiveness of the ProACTive intervention will be examined through scores on four standardised self-report measures of:

* Appearance concerns
* Positive and negative affect
* Psychological flexibility
* Self-compassion

These measures will be completed before and after the intervention. Wilcoxon tests will be used to compare pre- and post-intervention scores. These exploratory analyses will indicate the extent to which appearance concerns decrease, and psychological flexibility and self-compassion increase post-intervention compared to pre-intervention. Differences between pre- and post-intervention means will also give an indication of the likely effect size of the intervention (Cohen's d).

The outcome of the study will include knowledge about whether ProACTive is acceptable to burns patients when it is introduced during hospital admission and preliminary evidence about the effectiveness of ProACTive. These outcomes will contribute to further intervention refinement and trial development.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years and over) admitted as inpatients to the burns service with an acute burn injury

Exclusion Criteria:

* Patients already receiving psychological input from the burns clinical psychology service for appearance related concerns, over and above supportive listening
* Patients admitted as inpatients to the burns service for reconstructive surgery, for a historical burn injury
* Patients who are too physically unwell to participate
* Patients deemed too psychologically unwell or in a mental health crisis by the usual clinical care team (for example, patients who sustained their burn injury due to a suicide attempt or self-harm, are currently having suicidal thoughts, or those with psychosis)
* Patients who are not fluent in the English language in order to participate
* Patients with a known cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2024-06-13 (Actual); Primary Completion 2025-03-05 (Actual); Study Completion 2025-03-05 (Actual)

PRIMARY OUTCOMES:
Body Esteem Scale for Adolescents and Adults - Appearance subscale (BESAA-A) | As soon as is feasible before and after the intervention. The post-intervention measure will be completed within one week of the intervention ending
  A 10-item self-report questionnaire that measures appearance concerns/body esteem. Responses to each item fall on a scale between 0 and 4. The total mean score is used, falling between 0 and 4. Higher scores indicate higher appearance esteem (i.e. lower appearance concerns).

SECONDARY OUTCOMES:
Positive and Negative Affect Schedule (PANAS-GEN) | As soon as is feasible before and after the intervention. The post-intervention measure will be completed within one week of the intervention ending
  A 20-item standardised measure of positive and negative affect. Responses to items are scored between 1 and 5. Ten items relate to positive affect and 10 items relate to negative affect. Scores range from 10 to 50 for both sets of items. For the total positive score, a higher score indicates more positive affect. For the total negative score, a lower score indicates less negative affect. The total score is calculated by the sum of the 10 positive items and then the 10 negative items.
Comprehensive assessment of Acceptance and Commitment Therapy processes (CompACT) | As soon as is feasible before and after the intervention. The post-intervention measure will be completed within one week of the intervention ending
  A 23-item self-report questionnaire that measures psychological flexibility. Responses to each item fall on a scale between 0 and 6. The total score is used, ranging from 0 to 138. Three subscale scores can also be generated. Higher scores indicate greater psychological flexibility.
Self-Compassion Scale - Short Form (SCS-SF) | As soon as is feasible before and after the intervention. The post-intervention measure will be completed within one week of the intervention ending
  A 12-item self-report questionnaire that measures self-compassion. Responses to items fall on a scale between 1 and 5. The total mean score is used, with values ranging between 1 and 5. Higher scores indicate higher self-compassion.
Helpful Aspects of Therapy Form (HAT) | As soon as is feasible before and after the intervention. The post-intervention measure will be completed within one week of the intervention ending
  A seven-item self-report questionnaire that gathers mainly qualitative data about helpful and hindering aspects of therapy sessions.

CONTACTS AND LOCATIONS:
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Open Science Framework. Final template of themes (qualitative data).
Supporting Information: Study Protocol
Time Frame: Acceptance of manuscript for publication.
Access Criteria: The data will be made publicly available on the Open Science Framework upon acceptance of the manuscript for publication.

REFERENCES:
- [Background] Mendelson BK, Mendelson MJ, White DR. Body-esteem scale for adolescents and adults. J Pers Assess. 2001 Feb;76(1):90-106. doi: 10.1207/S15327752JPA7601_6. PMID 11206302
- [Background] Raes F, Pommier E, Neff KD, Van Gucht D. Construction and factorial validation of a short form of the Self-Compassion Scale. Clin Psychol Psychother. 2011 May-Jun;18(3):250-5. doi: 10.1002/cpp.702. Epub 2010 Jun 8. PMID 21584907
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Llewelyn SP. Psychological therapy as viewed by clients and therapists. Br J Clin Psychol. 1988 Sep;27(3):223-37. doi: 10.1111/j.2044-8260.1988.tb00779.x. PMID 3191302
- [Background] Francis, A. W., Dawson, D. L., & Golijani-Moghaddam, N. (2016). The development and validation of the Comprehensive Assessment of Acceptance and Commitment Therapy processes (CompACT). Journal of Contextual Behavioral Science, 5(3), 134-145.